CLINICAL TRIAL: NCT01773447
Title: Comparing Wound Eversion and Clinical Outcomes in Surgical Wound Repair With Subcuticular Set-back Versus Traditional Vertical Mattress Suturing Techniques
Brief Title: Set-back Suture Versus Traditional Vertical Mattress Suture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 247354
Record Dates: First submitted 2013-01-15; First posted 2013-01-23 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma; Melanoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Set-back suture (Active Comparator): Wound to be close by set-back suture technique.
  Interventions: Procedure: Set-back suture
- Vertical mattress suture technique (Active Comparator): Wound to be closed by vertical mattress technique.
  Interventions: Procedure: Vertical mattress suture

INTERVENTIONS:
Procedure: Set-back suture
  Arms: Set-back suture
Procedure: Vertical mattress suture
  Arms: Vertical mattress suture technique

SUMMARY:
The investigators hope to compare two different methods of closing skin wounds using sutures. One of these methods (the set-back technique) was recently described in 2010 and has been reported to be technically easier and reduces the chance of spitting sutures (deep sutures that are pushed to the surface of the skin as the wound heals). The other method (the vertical mattress technique) has been used for many years with good results. However, no controlled studies have been performed to clearly demonstrate a difference between the two methods. We hope to find differences in the height of the wound edges immediately after surgery(5 minutes following the procedure) as well as the appearance of the scar and symptoms associated with the scar 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elliptical surgical wound that needs to be closed with a layered closure
* Wound 3 cm in length or longer

Exclusion Criteria:

* Incarceration
* Active pregnancy
* Less than 18 years of age
* Unable to give informed consent
* Non-English or Dutch speaking (the scar assessment scale described below has only been validated in the English and Dutch languages)
* Wound closure projected to be less than 3 cm in length
* Skin less than 3 mm in thickness (dermis and epidermis combined)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Mean of sum of 2 blinded reviewers Physician Observer Assessment scores | 3 months
  Compare the functional and cosmetic outcomes of the two sutured halves of each scar at 3 months follow-up as follows:
  a. Use a previously validated scar assessment scale called the Patient and Observer Scar Assessment Scale, specifically the averaged sum of the total score of 2 blinded observers.
Scar width | 3 months
  Width of scar in millimeters for each side of scar measured 1 cm from the midline.

SECONDARY OUTCOMES:
Height of scar immediately following wound closure | 5 minutes
  Height of each side of the wound will be measured 1 cm from the midpoint of the wound in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis, Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical